CLINICAL TRIAL: NCT07370441
Title: A Single-Center, Prospective, Open-Label, Self-Controlled Clinical Study on the Efficacy and Safety of Amino Acid (15) Peritoneal Dialysis Solution in Improving Nutritional Status in Peritoneal Dialysis Patients
Brief Title: Amino Acid (15) Peritoneal Dialysis Solution for Nutritional Improvement in Peritoneal Dialysis Patients
Acronym: AA15-PD-Nut-SH
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Wen Xue MD, PhD, Attending Physician, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SH10H-AA15-PD-Nutrition
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: End-stage Renal Disease (ESRD); Peritoneal Dialysis (PD); Nutritional Status; Renal Replacement Therapy
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Amino Acids; Dialysis Solutions

STUDY DESIGN:
Intervention Model Description: This is a single-arm study with a self-controlled before-and-after design and no grouping. All participants will receive a uniform intervention: Amino Acid (15) Peritoneal Dialysis Solution replacement therapy, administered at a regular dose of 2L per session, once daily after lunch.
  The study will compare each participant's baseline health indicators (collected on the enrollment day) with those measured after 6 months of intervention to evaluate the efficacy and short-term safety of the intervention. No control group is included, as the comparison is conducted within the same participants to eliminate inter-individual confounding factors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amino Acid (15) PD Solution for Nutritional Support (Experimental): All participants will receive a uniform intervention: Amino Acid (15) Peritoneal Dialysis Solution replacement therapy, administered at a regular dose of 2L per session, once daily after lunch.
  Interventions: Drug: amino acid (15) peritoneal dialysis solution

INTERVENTIONS:
Drug: amino acid (15) peritoneal dialysis solution — Amino Acid (15) Peritoneal Dialysis Solution replacement therapy, administered at a regular dose of 2L per session, once daily after lunch.

SUMMARY:
The goal of this clinical trial is to assess whether Amino Acid (15) Peritoneal Dialysis Solution can improve the nutritional status of adults with end-stage kidney disease who have received peritoneal dialysis for 6 months or longer. It will also observe the solution's effects on dialysis adequacy and peritoneal transport function, as well as monitor its short-term safety. The main questions it aims to answer are:

1. Can Amino Acid (15) Peritoneal Dialysis Solution raise the level of serum albumin (a key indicator of nutritional status) in participants?
2. How does this solution affect participants' dialysis adequacy and peritoneal transport function?
3. What adverse reactions might participants experience when using this solution? This is a single-arm study with a self-controlled design. Researchers will compare participants' health indicators before and after the intervention to evaluate the solution's effectiveness and safety.

Participants will:

1. Continue their original peritoneal dialysis routine, replacing one bag of dialysis solution with Amino Acid (15) Peritoneal Dialysis Solution (2L per bag) after lunch every day for 6 months.
2. Undergo comprehensive health checks (including blood tests, nutritional status assessments, and peritoneal function evaluations) on the enrollment day (baseline), as well as at 3 and 6 months after the intervention.
3. Attend follow-up visits every 2 weeks to record dialysis-related data (such as ultrafiltration volume) and any uncomfortable symptoms or adverse reactions.
4. Maintain stable doses of medications affecting protein metabolism and nutritional supplements throughout the study; report to researchers immediately if any dose

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Have received peritoneal dialysis for 6 months or longer.
3. Serum albumin level < 38 g/L.
4. No history of peritonitis in the past 3 months and no hospitalization in the past 1 month.
5. No severe heart, liver, kidney diseases, or malignant tumors.
6. Expected survival time > 1 year.
7. Good compliance and willingness to sign the informed consent form.
8. Diagnosed with end-stage renal disease (ESRD) with an estimated glomerular filtration rate (eGFR) < 15 mL/(min·1.73 m²).

Exclusion Criteria:

1. Hypersensitivity or allergy to Amino Acid (15) Peritoneal Dialysis Solution or any of its components.
2. Hepatic dysfunction (ALT/AST ≥ 2 times the upper limit of normal).
3. Taking medications that affect protein metabolism and unable to maintain a stable dose during the study period.
4. Need for adjustment of nutritional supplement doses during the study.
5. Uncorrectable severe gastrointestinal reactions.
6. Pregnant, lactating, or planning to undergo kidney transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum Albumin (Alb) | At baseline (enrollment day), at 3 months into the intervention, and at the end of the 6-month intervention period

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-12-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT07370441/Prot_ICF_000.pdf